CLINICAL TRIAL: NCT02851615
Title: SCThrive: Improving Self-Management in Adolescents With Sickle Cell Disease
Brief Title: Improving Self-Management in Adolescents With Sickle Cell Disease
Acronym: SCThrive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21HD084810-01A1 (NIH)
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Sickle Cell Disease
Keywords: Anemia, Sickle Cell; Self Care; Adolescent; Young Adult; Disease Management; Behavioral Activation; Peer Communication
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCThrive (Other): SCThrive Intervention for Adolescents with SCD - 6 week self-management group
  Interventions: Behavioral: SCThrive Intervention for Adolescents with SCD
- Attention Control (No Intervention): 6 weekly 15-20 minute individual phone calls on educational topics. No interventions are included in this arm.

INTERVENTIONS:
Behavioral: SCThrive Intervention for Adolescents with SCD — Chronic Disease Self-Management Program
  Arms: SCThrive

SUMMARY:
The objective of this study is to determine the feasibility and acceptability of SCThrive, a an innovative, technology-enhanced, group self-management intervention that uses a mixed in-person and online format and supported by a tailored mHealth tool, iManage. The study will also evaluate the initial efficacy of SCThrive for increasing behavioral activation (BA) in adolescents with Sickle Cell Disease (SCD) ages 13 to 21. The investigators hypothesize that participants in the SCThrive group will show greater BA (primary outcome) at post-treatment than the attention control group, and that participants in the SCThrive group will continue to show significantly greater BA at the six week follow-up compared to the attention control group. Investigators will also explore whether SCThrive is associated with greater improvements in self-management behaviors and quality of life (secondary outcome) compared to attention control at the six-week follow-up assessment.

DETAILED DESCRIPTION:
The objective of this study is to determine the feasibility and acceptability of SCThrive, a an innovative, technology-enhanced, group self-management intervention that uses a mixed in-person and online format and supported by a tailored mHealth tool, iManage. The study will also evaluate the initial efficacy of SCThrive for increasing behavioral activation (BA) in adolescents with Sickle Cell Disease (SCD) ages 13 to 21.

ELIGIBILITY:
Inclusion Criteria:

* Patient of CCHMC Sickle Cell Clinic.
* Confirmed diagnosis of SCD with SS, SB0Thal or SC genotype.
* 13-21 years of age.
* On or eligible for disease-modifying therapies.
* Caregiver (or AYA > 18 years) consent that the participant will be the sole user of the tablet, report immediately if it is damaged or lost, return it at the end of the study, and log on to sessions from a private location.

Exclusion Criteria:

* another chronic disease (which would complicate measurement of behavioral activation)
* Non-English-speaking (<5% of the target population); or
* cognitive or psychiatric disorder that the physician or study therapists believe would impair study participation. Patients who desire participation but are not eligible will be referred to the SCD Clinic social worker for assistance with self-management as this is the usual procedure.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori E Crosby, PsyD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crosby LE, Modi AC, Lemanek KL, Guilfoyle SM, Kalinyak KA, Mitchell MJ. Perceived barriers to clinic appointments for adolescents with sickle cell disease. J Pediatr Hematol Oncol. 2009 Aug;31(8):571-6. doi: 10.1097/MPH.0b013e3181acd889. PMID 19636266
- [Background] Crosby LE, Joffe NE, Reynolds N, Peugh JL, Manegold E, Pai AL. Psychometric Properties of the Psychosocial Assessment Tool-General in Adolescents and Young Adults With Sickle Cell Disease. J Pediatr Psychol. 2016 May;41(4):397-405. doi: 10.1093/jpepsy/jsv073. Epub 2015 Aug 13. PMID 26275975
- [Background] Crosby LE, Joffe NE, Dunseath LA, Lee R. Design Joins the Battle Against Sickle-cell Disease. Des Manage Rev. 2013 Summer;24(2):48-53. doi: 10.1111/drev.10241. No abstract available. PMID 25414599
- [Result] Crosby LE, Hood A, Kidwell K, Nwankwo C, Peugh J, Strong H, Quinn C, Britto MT. Improving self-management in adolescents with sickle cell disease. Pediatr Blood Cancer. 2020 Oct;67(10):e28492. doi: 10.1002/pbc.28492. Epub 2020 Jul 22. PMID 32697889

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SCThrive | Attention Control
Started | 27 | 31
Completed | 26 | 27
Not Completed | 1 | 4
Not completed — Cognitive Issue | 1 | 0
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCThrive | Attention Control | Total
Number analyzed (Participants) | 27 | 31 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant in SC Thrive did not complete the intervention due to a cognitive issue (n=1).
  Four participants in Attention Control did not complete the intervention and were lost to follow-up (n=4).
  years
    number analyzed (Participants) | 26 | 27 | 53
    (all) | 16.7 (2.3) | 16.3 (2.5) | 16.5 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant in SC Thrive did not complete the intervention due to a cognitive issue (n=1).
  Four participants in Attention Control did not complete the intervention and were lost to follow-up (n=4).
  Participants
    number analyzed (Participants) | 26 | 27 | 53
    Female | 14 | 14 | 28
    Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant in SC Thrive did not complete the intervention due to a cognitive issue (n=1).
  Four participants in Attention Control did not complete the intervention and were lost to follow-up (n=4).
  Participants
    number analyzed (Participants) | 26 | 27 | 53
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 26 | 27 | 53
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant in SC Thrive did not complete the intervention due to a cognitive issue (n=1).
  Four participants in Attention Control did not complete the intervention and were lost to follow-up (n=4).
  Participants
    number analyzed (Participants) | 26 | 27 | 53
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 26 | 27 | 53
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 31 | 58

OUTCOME MEASURES:

1. Primary Outcome: Scores on Behavioral Activation Measure at Baseline and 6 Weeks (Post-treatment)
Description: Participants complete the Patient Activation Measure (PAM-13), which is a 13 item measure on skills, knowledge, confidence and readiness for self-management developed by Hibbard et al., 2005. Items are rated on a 4-point Likert scale of 1 = "Disagree Strongly" to 3 = "Strongly Agree." Raw scores range from 13 to 52 and are converted to scores that range from 0 to 100. This score was then divided into four levels of activation, which reflect a developmental progression from being passive with regard to one's health to being proactive: Level 1 (score of 0.0 - 47.0), Level 2 (47.1 - 55.1), Level 3 (55.2 - 72.4), and Level 4 (72.5 - 100). Higher scores indicate more behavioral activation.
Time Frame: baseline, 6 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCThrive | Attention Control
Number analyzed (Participants) | 26 | 27
score on a scale
  Baseline Scores | 68.48 (15.47) | 69.13 (20.75)
  Post- Treatment Scores | 76.57 (15.04) | 68.82 (18.18)
Statistical Analysis 1: Comparison: SCThrive vs Attention Control; We conducted separate mixed ANOVA analyses to assess for the effects of group (SCThrive/SCHealthEd), time (baseline/post-treatment), and group x time interaction for the PAM-13; Test type: Superiority — Power analyses were calculated on the PAM-13, our primary outcome measure. Analyses were conducted using the internal Monte Carlo simulation capabilities of Mplus (Version 1.20). Based on the effect size obtained from published pilot data, we expected the change in baseline/posttreatment Behavioral Activation for the SCThrive intervention group to be n2 = .14 (large effect). Based on these assumptions, the desired sample size was 54 participants (N = 27 per group) to achieve power of .80; p = .09, ANCOVA — The threshold for statistical significance was p =.05; Mean Difference (Net) = 7.75, 95% CI 2-sided [-1.27 to 19.22], Standard Error of Mean 13.14

2. Secondary Outcome: Scores on a Self-management Measure at Baseline and 6 Weeks (Post-treatment)
Description: Participants complete the Transition Readiness Assessment Questionnaire (TRAQ-5), which is a well-validated 20-item questionnaire that measures the skills needed to manage a chronic condition independently. Items are rated on a 5-point Likert scale of 1 = "No, I do not know how" to 5 = "Yes, I always do this when I need to" and divided into 5 subscales: Managing Medication, Appointment Keeping, Tracking Health Issues, Talking with Providers, and Managing Daily Activities. Overall and subscale scores are calculated by averaging the scores of answered items. Mean scores range from 1 to 5 with higher scores indicating better self-management.
Time Frame: baseline, 6 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCThrive | Attention Control
Number analyzed (Participants) | 26 | 27
score on a scale
  Baseline Scores | 3.46 (.83) | 3.54 (.81)
  Post-Treatment Scores | 3.68 (.81) | 3.53 (.79)
Statistical Analysis 1: Comparison: SCThrive vs Attention Control; We conducted separate mixed ANOVA analyses to assess for the effects of group (SCThrive/SCHealthEd), time (baseline/post-treatment), and group x time interaction for the TRAQ-5; Test type: Superiority; p = .28, ANCOVA — The threshold for significance was p =.05; Mean Difference (Net) = .15, 95% CI 2-sided [-.19 to .66], Standard Error of Mean .55

3. Secondary Outcome: Total Scores on the UNC TRxANSITION Scale at Baseline and 6 Weeks Post-Treatment
Description: Participants complete the UNC TRxANSITION Scale, an interview administered by trained independent evaluators to measure the skills of youth with chronic conditions. For this study, we administered 6 of the 10 possible subscales: Type of Chronic Health Condition, Medications, Adherence, Nutrition, Self-Management Skills, and New Health Care Providers. Each item is scored individually as either 1 (adequate knowledge/skill mastery), 0.5 (some knowledge/skill attainment), or 0 (no knowledge/skill attainment). Higher scores indicate better self-management. Subscale scores are calculated by dividing the patient's score by the total possible subscale score. Subscale scores are then combined to create a total score, ranging from 0 to 10, but since we only used 6 scales, 0 to 6. Total and subscale proportion scores were used in analyses.
Time Frame: baseline, 6 weeks (post-treatment)
Population: Data assessing transition readiness (UNC TRxANSITION Scale) were only collected from adolescents and and young adults completing SCThrive (N=16).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SCThrive: SCThrive Intervention for Adolescents with SCD - 6-week self-management group
Arm/Group | SCThrive
Number analyzed (Participants) | 16
score on a scale
  Baseline Score | 1.19 (.13)
  Post-Treatment Score | 1.15 (.11)
Statistical Analysis 1: Comparison: SCThrive; We conducted a paired-samples t-test to assess for the effects of time (baseline/post-treatment) for participants (n=16) in the SCThrive intervention arm for the UNC TRxANSITION Scale; Test type: Superiority; p = .27, t-test, 2 sided — The threshold for statistical significance was p =.05; Mean Difference (Net) = .02, 95% CI 2-sided [-.018 to .06], Standard Deviation .13

ADVERSE EVENTS:
Time Frame: baseline, 6 weeks (post-treatment)
Description: Monthly meetings to monitor the progress of the study, the integrity of the treatment and safety monitoring, including a review of any adverse events. If adverse events, investigators followed-up and provided referral or treatment until the event subsided. Investigators were available 24 hours via pager. The PI reported any significant study-related or unanticipated adverse events to the Institutional Review Board and study sponsor based upon institutional and sponsor guidelines.
Arm/Group | SCThrive | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT02851615/Prot_SAP_000.pdf